CLINICAL TRIAL: NCT05486650
Title: An Observational Clinical Study of Increasing Stereotactic Radiotherapy in Patients With Advanced Non-small Cell Lung Cancer After Treatment With PD-1 Inhibitors And Evaluation of Stable Disease
Brief Title: An Observational Clinical Study of Stereotactic Radiotherapy for Advanced Non-Small Cell Lung Cancer With Stable Disease After PD-1 Inhibitor Treatment
Status: Recruiting | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Chief physician, Xinqiao Hospital of Chongqing
Other Study IDs: 2021-yandi147-01
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors; Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PD-1 inhibitor — After receiving PD-1 inhibitor treatment in the first three cycles, patients with locally advanced or advanced NSCLC whose curative effect is evaluated as stable disease receive SBRT combined with PD-1 inhibitor treatment
  Other Names: Stereotactic Body Radiation Therapy

SUMMARY:
After the treatment of advanced non-small cell lung cancer with immune checkpoint inhibitor PD-1/PD-L1 monoclonal antibody, if the treatment response of complete response (CR) or partial response (PR) can be achieved in the early stage, the patients are expected to obtain a better long-term survival rate. Radiotherapy can synergistically improve the effect of immunotherapy. Therefore, we propose a hypothesis: in patients with advanced lung cancer, if only stable disease (SD) is achieved after PD-1 antibody immunotherapy in the early stage, by increasing the stereotactic radiotherapy (SBRT) for primary or metastatic lesions, in order to improve the mechanism of tumor antigen release, promote the activation and activation of effector T cells, and increase the sensitivity of immunotherapy, so as to achieve the goal of early improvement of objective remission rate (ORR). It is expected to improve the long-term survival rate of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed, and according to the judgment of the investigator, the patient can comply with the study protocol;
2. Patients with stage IIIB, IIIC and stage IV NSCLC (according to the definition of the 8th edition of the American Joint Commission on cancer), who have not been treated and cannot receive radical surgery or radiotherapy confirmed by histopathology, received 3-4 cycles of PD1 antibody ± chemotherapy in the early stage, and the efficacy was evaluated as SD;
3. Previously, no EGFR sensitive mutation and ALK, ROS1 gene fusion mutation were detected based on tissue examination;
4. There are measurable lesions evaluated by researchers according to RECIST version 1.1;
5. The physical state score (ECOG PS) of the eastern cancer cooperation group was 0-1;
6. Good cardiopulmonary function

Exclusion Criteria:

1. The patient's compliance is poor and violates the test regulations;
2. Patients with positive driver gene are known to carry EGFR mutation or ALK, ROS1 gene translocation;
3. There are dysfunction of important organs of liver and kidney, such as myocardial infarction, angina pectoris, liver transaminase significantly increased;
4. Serious adverse drug reactions occurred during induction;
5. Have suffered from any disease requiring systemic treatment with corticosteroids or other immunosuppressive drugs within 14 days before enrollment;
6. Severe infection occurred within 4 weeks before enrollment, including but not limited to hospitalization due to infection complications, bacteremia or severe pneumonia;
7. Severe chronic or active infection (including tuberculosis infection) requiring systemic (oral or intravenous) antibiotic treatment within 14 days before enrollment;
8. Have a history of interstitial lung disease, non infectious pneumonia or poorly controlled diseases, including pulmonary fibrosis, acute lung disease, etc;
9. Untreated patients with chronic hepatitis B, HBV carriers with hepatitis B virus (HBV) DNA ≥ 500 iu/ml, or patients with active hepatitis C virus (HCV) should be excluded;
10. Known history of HIV infection;
11. Received any other trial drug treatment or participated in other clinical trials within 28 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage IIIB, IIIC and stage IV NSCLC (according to the definition of the 8th edition of the American Joint Commission on cancer), who have not been treated and cannot receive radical surgery or radiotherapy confirmed by histopathology, received 3-4 cycles of PD1 antibody ± chemotherapy in the early stage, and the efficacy was evaluated as stable disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 2 year
  The proportion of patients whose tumors shrink to a certain amount and remain for a certain period of time, including cases of complete response and partial response.

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality, China